CLINICAL TRIAL: NCT06832904
Title: Neoadjuvant Chemotherapy Plus Pyrotinib and Trastuzumab for HER2-positive Breast Cancer (NEOTORCH-BREAST05): A Prospective, Single-arm, Multi-center Clinical Study
Brief Title: Neoadjuvant Chemotherapy Plus Pyrotinib and Trastuzumab for HER2-positive Breast Cancer (NEOTORCH-BREAST05)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20240161C-R1
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-12

CONDITIONS: HER2-positive Breast Cancer; Neoadjuvant Therapy; Pyrotinib
MeSH Terms: interventions — pyrotinib; Trastuzumab; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single-arm (Experimental)
  Interventions: Drug: pyrotinib and trastuzumab in combinition with neoadjuvant chemotherapy

INTERVENTIONS:
Drug: pyrotinib and trastuzumab in combinition with neoadjuvant chemotherapy — Receive four neoadjuvant cycles of oral pyrotinib (400 mg) once daily, plus intravenous trastuzumab (8 mg/kg loading dose, followed by 6 mg/kg) , nab-paclitaxel (260 mg/m2) and carboplatin（AUC=5）every 3 weeks.

SUMMARY:
This study is a prospective, single arm, multi-center clinical trial. The primary study objective is to evaluate the pathologic complete response (pCR）and clinical complete response（cCR) of neodjuvant treatment of HER2-positive breast cancer with pyrotinib and trastumab combined with neoadjuvant chemotherapy. The secondary study objective is to observe and evaluate the disease-free survival (DFS), Progression-Free-Survival (PFS ),and Objective Response Rate(ORR). The study also observes the incidence and types of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18-75 years old; 2. ECOG score is 0-1 points; 3. Histologically confirmed invasive cancer meets the following standards:

* T1N1-3M0 or T2-4N0M0
* All patients were pathohistologically confirmed as HER2+ breast cancer. HER2 positivity was determined locally and defned as 3+ staining intensity by immunohistochemistry or HER2 gene amplifcation by fuorescence in situ hybridization according to the 2013 American Society of Clinical Oncology/College of American Pathologists guidelines.

  4. The functional level of major organs must meet the following requirements (no blood transfusion, no use of leukocyte and platelet boosting drugs within 2 weeks before screening):
  1. Blood routine: Absolute neutrophil count (ANC) greater than 1.5 × 109/L; platelet count (PLT) greater than 75 × 109/L; Hemoglobin (Hb) is greater than 90g/L; Lymphocyte count ≥ 1.5 × 109/L
  2. Blood biochemistry: Total bilirubin (TBIL) is less than 1.5 × ULN; Alanine aminotransferase (ALT) and aspartate (AST) levels are less than 1.5 × ULN; Alkaline phosphatase is less than 2.5 × ULN; Urea nitrogen/Urea (BUN/UREA) and creatinine (Cr) are less than 1.5 × ULN.
  3. Cardiac ultrasound: Left ventricular ejection fraction (LVEF) greater than 55%.
  4. 12 lead electrocardiogram: The Fridericia corrected QT interval (QTcF) is less than 470 milliseconds 5. For female patients who have not yet reached menopause or undergone surgical sterilization: during the treatment period and in the study treatment, the final use effective contraceptive methods for at least 6 months after a single administration.

  6. Voluntarily join this study, sign an informed consent form, have good compliance, and are willing to cooperate with follow-up.

Exclusion Criteria:

1. Stage IV breast cancer.
2. Inflammatory breast cancer.
3. Previously received anti-tumor treatment or radiation therapy for any malignant tumor, excluding those that have been cured malignant tumors such as cervical carcinoma in situ, basal cell carcinoma, or squamous cell carcinoma.
4. Simultaneously undergoing anti-tumor treatment in other clinical trials, including but not limited to chemotherapy, endocrine therapy, biological therapy, bone improvement drug therapy, or immune checkpoint inhibitor therapy, etc.
5. The patient had undergone major surgical procedures unrelated to breast cancer within 4 weeks before the first administration of the study drug, or the patient has not fully recovered from such surgical procedures.
6. Serious heart disease or discomfort, including but not limited to the following diseases:

1) Diagnosed history of heart failure or systolic dysfunction (LVEF less than 50%).

2) High risk uncontrolled arrhythmias, such as atrial tachycardia, resting heart rate greater than 100bpm, significant ventricular arrhythmias (such as ventricular tachycardia), or higher-level atrioventricular block (i.e. Mobitz II second or third degree atrioventricular block).

3) Angina requiring medication for treatment. 4) Heart valve disease with clinical significance. 5) ECG shows transmural myocardial infarction. 6) Poor control of hypertension (systolic blood pressure greater than 180mmHg and/or diastolic blood pressure greater than 100mmHg after drug treatment).

7. Uncontrolled active infections that require treatment; History of immunodeficiency, including HIV testing positive Sexual, or suffering from other acquired or congenital immunodeficiency diseases, or having a history of organ transplantation.

8. Patients with chronic active hepatitis B or active hepatitis C (excluding hepatitis B virus carriers, stable hepatitis B after drug treatment [HBV-DNA test negative or<50IU/ml] and cured hepatitis C patients [HCV RNA test negative]).

9. Individuals with a known history of allergies to the components of this medication regimen.

10. Pregnant and lactating female patients, female patients with fertility and positive baseline pregnancy test results, or reproductive age patients who are unwilling to take effective contraceptive measures during the entire trial period and within 6 months after the last study medication.

11. Suffering from serious accompanying diseases or other comorbidities that may interfere with the planned treatment, or any other circumstances that the researcher deems unsuitable for the patient to participate in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response（pCR） | 2 years
clinical complete response（cCR) | 2 years

SECONDARY OUTCOMES:
RCB 0-1 ratio | 2 years
disease-free survival (DFS) | 3 years
progression-free survival (PFS) | 3 years
objective response rate (ORR) | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, China